CLINICAL TRIAL: NCT00977158
Title: Microbiota of the Respiratory Flora in Children With Cystic Fibrosis During the First Year of Life
Status: Withdrawn | Type: Observational
Why Stopped: No problems with planned study- insufficient funding for this study to proceed.
Sponsor: Tufts Medical Center (Other)
Responsible Party: Patricia L. Hibberd, MD, PhD, Tufts Medical Center
Other Study IDs: 8851
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Microbiota; upper respiratory tract; 16S rRNA sequence analysis; Staphylococcus aureus; Pseudomonas aeruginosa; Burkholderia cepacia; Haemophilus influenzae; Streptococcus pneumoniae
MeSH Terms: conditions — Cystic Fibrosis; Staphylococcal Infections; Pseudomonas Infections; Haemophilus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Throat Swab: Infants who have been diagnosed with cystic fibrosis
  Interventions: Procedure: Throat Swab

INTERVENTIONS:
Procedure: Throat Swab — Swabs will be moistened in sterile 0.9% sodium chloride solution and rotated in the throat and processed for bacterial cultures and for bacterial DNA extraction.

SUMMARY:
The goal of this study is characterize the changes in bacterial diversity of the upper respiratory tracts of infants with cystic fibrosis (CF). Another goal is to determine when CF patients become colonized with pathogenic bacteria that are responsible for the lethal lung damage in children with CF. Ten subjects will be recruited into the study. Throat swabs will be collected at 6-8 weeks of age, 3 months, 6 months, 9 months, and 12 months of age in order to chart any changes in the bacterial populations of the respiratory tract. Clinical data will also be collected to evaluate the possible influence of external factors on changes in the microbial communities. This study will provide preliminary data on whether probiotics can eradicate the colonization of the respiratory tract by pathogenic bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, newborn to age 3 months
* Have a diagnosis of cystic fibrosis (Diagnosis of CF will be based on either a positive sweat chloride of >60 mEq/L or the identification of two detectable mutations associated with CF
* Parent/guardian plans to have follow-up care for approximately one year at designated CF clinic
* Parent/guardian provides informed consent to participate in the study

Exclusion Criteria:

* Contraindications for obtaining oropharyngeal swabs

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-05

PRIMARY OUTCOMES:
To characterize the microbial ecology and changes in bacterial diversity of the oropharynx in a cohort of children with CF during the first year of life using 16S rRNA sequence analysis | 6-8 weeks of age, 3 months, 6 months, 9 months, and 12 months of age
To describe the clinical variables that may be associated with changes in microbial ecology in children with cystic fibrosis over the first year of life | 6-8 weeks of age, 3 months, 6 months, 9 months, and 12 months of age
To explore changes in the microbial ecology of the oropharynx in conjunction with Staphylococcus aureus colonization in children with CF | 6-8 weeks of age, 3 months, 6 months, 9 months, and 12 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L Hibberd, MD, PhD, Principal Investigator — Tufts Medical Center
Locations (2):
- United States (2):
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts